CLINICAL TRIAL: NCT04382742
Title: Exercise Response on Dose Curve Among Class I Obese Young Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Batool Hassan, Principal Investigator, Ziauddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BatoolH
Record Dates: First submitted 2020-05-01; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental)
  Interventions: Behavioral: Dynamic Resistance Exercises

INTERVENTIONS:
Behavioral: Dynamic Resistance Exercises — Modified Wingate protocol that incorprates 20 minutes of training on a cycle ergometer; included one minute of cycling with resistance to be performed at 85% to 90% of Maximal Heart Rate (MHR) followed by one minute of cycling with no resistance. The protocol will be performed for 10 times for a duration of 20 minute of workout.

SUMMARY:
The study is aimed to determine impact of dynamic resistance exercise training on Body Fat percentage of class-I Obese population and to quantify the dose of exercise program using a probit regression curve

DETAILED DESCRIPTION:
Methodology

A sample size of 34 participants 17 male and 17 female of aged between 20-40 years with class-I obesity were selected and recruited in this study. All the participants were initially screened using a physical activity and readiness questionnaire to determine if they are fit to perform exercises afterwards intervention based on dynamic exercises were given to the patient for 12 weeks based on the guidelines of American College of Sports Medicine and the quantification of exercises was done using a Frequency, Intensity, Time and Type (FITT) protocol. The training session was based on Warm up 5 to 10 minutes followed by conditioning phase of 20 minutes and a cool down phase of 5 to 10 minutes. The detailed description of each of the phase is as under:

Warm up Phase Dynamic light aerobic warm up exercises were performed by the participants for 5 to 10 minutes before the start of the conditioning. Two different exercises that were performed included i) High Knee in which the knees will be lifted as high as possible in such a manner that both feet should be at one time be above the ground ii) Jumping Jack Exercise in which a simultaneous movement of upper and lower limb will be performed in a manner that every time during a jump the arms were thrusted over the head while the foot moved out to the side and than returning back to the original position 10 repetitions of both the exercises were performed.

Dynamic Resistance Exercise Modified Wingate protocol that incorporates 20 minutes of training on a cycle ergometer; included one minute of cycling with resistance to be performed at 85% to 90% of Maximal Heart Rate (MHR) followed by one minute of cycling with no resistance. The protocol will be performed for 10 times for a duration of 20 minute of workout.

Cool Down The process of cool down last for 5-10 minutes. During this low intensity, long hold stretching were performed of lower limb and upper limb that included shoulder, calf and hamstring stretch

ELIGIBILITY:
Inclusion Criteria:

* • Class I obese population BMI 30 -39.9

  * Young adults of age 20-40 years
  * Male and female population

Exclusion Criteria:

* • Recent surgery that limits participation in exercise program

  * Known Cardia Disease
  * Any comorbidity that limits participation in training program

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage (Pre treatment) | Baseline
  Body fat percentage is used to measure fat mass with higher percentage revealing greater body fat. The values are calculated using skin fold thickness (precision caliper) method.
Body Fat Percentage (Post treatment) | After 12 weeks of training
  Body fat percentage is used to measure fat mass with higher percentage revealing greater body fat. The values are calculated using skin fold thickness (precision caliper) method.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No